CLINICAL TRIAL: NCT04581070
Title: COVID-IYON Study. Prospective, Multisite, Descriptive, Observational Clinical/Epidemiological Study Examining Data Pertaining to Clinical Outcomes and Organizational Responses to the 2020 SARS-Coronavirus-2 (SARS-CoV-2) Pandemic
Brief Title: The COVID-IYON Study - Study Examining Data Pertaining to Clinical Outcomes and Organisational Responses to the 2020 SARS-CoV-2 Pandemic"
Status: Terminated | Type: Observational
Why Stopped: Study stopped due to low accrual
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE 20-01
Record Dates: First submitted 2020-05-29; First posted 2020-10-09 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Cancer; COVID-19
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multisite, descriptive, observational clinical/epidemiological study examining both quantitative and qualitative data pertaining to clinical outcomes and organizational responses to the 2020 SARS-Coronavirus-2 (SARS-CoV-2) pandemic.

DETAILED DESCRIPTION:
This study collects real-time observational data regarding the impact of SARS-CoV-2 infection on patients with cancer, and on the functioning and organisation of cancer and malignant haematology services in the Republic of Ireland in response to the 2020 SARS-CoV-2 pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Informed consent has been obtained.
3. Cytotoxic chemotherapy, targeted anticancer therapy, immunomodulatory anticancer therapy, hormonotherapy, radiotherapy, oncologic surgery, or other anticancer treatment within the last 12 months (ongoing and completed).
4. Tested positive for SARS-CoV-2.

Exclusion Criteria:

There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of medical oncology & malignant haematology services, admitted at participating sites, who test positive for SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
A qualitative description | Up til 1 year
  A qualitative narrative description of national cancer care practises and risk mitigation strategies adopted in response to the SARS-CoV-2 pandemic.

CONTACTS AND LOCATIONS:
Locations (3):
- Ireland (3):
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: Undecided